CLINICAL TRIAL: NCT00454805
Title: A Phase II, Double-Blind, Placebo Controlled, Randomized Study to Assess the Efficacy and Safety of AZD2171 in Combination With Fulvestrant vs Fulvestrant Alone in Hormone Sensitive (ER+ve or PgR+ve) Post Menopausal Metastatic Breast Cancer Patients
Brief Title: AZD2171 in Addition to Fulvestrant in Patients With Advanced Breast Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D8480C00007
Record Dates: First submitted 2007-03-29; First posted 2007-04-02 (Estimated); Results first posted 2012-11-28 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-07

CONDITIONS: Advanced Breast Cancer
Keywords: Advanced Breast Cancer
MeSH Terms: interventions — cediranib; Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 2 (Active Comparator): Fulvestrant Monotherapy
  Interventions: Drug: Fulvestrant
- 3 (Experimental): AZD2171 + Fulvestrant
  Interventions: Drug: AZD2171; Drug: Fulvestrant

INTERVENTIONS:
Drug: AZD2171 — Oral tablet
  Other Names: Recentin
  Arms: 3
Drug: Fulvestrant — intramuscular injection
  Other Names: Faslodex; ZD9238

SUMMARY:
The purpose of this study is to determine whether AZD2171 can effectively improve time to tumour progression when added to fulvestrant in patients with advanced hormone sensitive breast cancer who progressed on prior hormonal therapy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Females with histological/cytological confirmation of hormone sensitive breast cancer with evidence of metastatic disease
* One or more evaluable lesions

Exclusion Criteria:

* Prior hormonal therapy with fulvestrant
* More than one course of prior systemic cytotoxic chemotherapy for metastatic breast cancer
* Prior biologic therapy for ABC including Anti-VEGF agents
* Radiation therapy within 4 weeks prior to provision of consent

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bijoyesh Mookerjee, MD, Study Director — AstraZeneca
Locations (16):
- United States (6):
  - Research Site, Burbank, California
  - Research Site, Los Angeles, California
  - Research Site, Palm Springs, California
  - Research Site, Boca Raton, Florida
  - Research Site, Honolulu, Hawaii
  - Research Site, New York, New York
- Australia (4):
  - Research Site, Fitzroy
  - Research Site, Parkville
  - Research Site, Perth
  - Research Site, Waratah
- Brazil (6):
  - Research Site, Belo Horizonte
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Porto Alegre
  - Research Site, Santro Andre
  - Research Site, São Paulo

REFERENCES:
- [Derived] Hyams DM, Chan A, de Oliveira C, Snyder R, Vinholes J, Audeh MW, Alencar VM, Lombard J, Mookerjee B, Xu J, Brown K, Klein P. Cediranib in combination with fulvestrant in hormone-sensitive metastatic breast cancer: a randomized Phase II study. Invest New Drugs. 2013 Oct;31(5):1345-54. doi: 10.1007/s10637-013-9991-2. Epub 2013 Jun 26. PMID 23801303
- See also: CSR-D8480C00007.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=416&filename=CSR-D8480C00007.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomised=ITT=Safety: Cediranib 31, Placebo 31
Pre-assignment Details: In this study, 75 patients were enrolled and 62 randomised.
Groups:
- Cediranib 45 mg: Cediranib 45 mg+Fulvestrant 250 mg
  Patients randomised to the investigational arm (fulvestrant + cediranib) received treatment according to the following schedule:
  * Day 1: fulvestrant 500 mg im
  * Day 15: fulvestrant 250 mg im
  * Day 29, and every 28 days thereafter: fulvestrant 250 mg im
  * and daily: cediranib 45 mg (administered orally)
- Placebo: Placebo+Fulvestrant 250 mg
  Patients randomised to the control arm (fulvestrant + placebo) received treatment according to the following schedule:
  * Day 1: fulvestrant 500 mg im
  * Day 15: fulvestrant 250 mg im
  * Day 29, and every 28 days thereafter: fulvestrant 250 mg im
  * and daily: placebo to match cediranib (administered orally)
Period: Overall Study
Arm/Group | Cediranib 45 mg | Placebo
Started | 31 (Randomised) | 31 (Randomised)
Completed | 5 (Ongoing at data cut-off) | 8 (Ongoing at data cut-off)
Not Completed | 26 | 23
Not completed — Withdrawal by Subject | 9 | 2
Not completed — Death | 0 | 2
Not completed — Disease progression | 16 | 19
Not completed — In order to begin radiotherapy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cediranib 45 mg | Placebo | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.4 (11.4) | 57.9 (9.7) | 59.1 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 31 | 62
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Number of months from randomisation until progressive disease based on RECIST (progression of target lesions, clear progression of existing non-target lesions or the appearance of one or more new lesions) or death in the absence of progression.
Time Frame: RECIST performed at screening and every 8 weeks through to progression or discontinuation whichever is earliest.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Cediranib 45 mg | Placebo
Number analyzed (Participants) | 31 | 31
Days | 223 [129 to 340] | 112 [59 to 329]

2. Secondary Outcome: Objective Response Rate
Description: Best objective tumour response (based on Response Evaluation Criteria in Solid Tumours (RECIST)) during the study for patients with measurable disease. Best objective tumour response defined as:
  Complete Response (CR) Disappearance of all target lesions Partial response (PR) At least a 30% decrease in the sum of longest diameters (LDs) of target lesions, taking as reference the baseline sum of LDs.
  Progression (PD) At least a 20% increase in the sum of LDs of target lesions, taking as reference the smallest sum of LDs since treatment started (including the baseline sum of LDs) and at least 5 mm increase.
  Stable disease (SD) Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD
Time Frame: RECIST performed at screening and every 8 weeks through to progression or discontinuation whichever is earliest.
Measure: Number; unit: Participants
Arm/Group | Cediranib 45 mg | Placebo
Number analyzed (Participants) | 18 | 12
Participants | 4 | 1

3. Secondary Outcome: Duration of Response
Description: Number of days from date of response (complete/partial based on RECIST) to date of progression
Time Frame: Every 8 weeks until progression or discontinuation
Measure: Median (Full Range); unit: Days
Arm/Group | Cediranib 45 mg | Placebo
Number analyzed (Participants) | 31 | 31
Days | 207.5 [82 to 396] | 224.0 [224 to 224]

4. Secondary Outcome: Clinical Benefit Rate
Description: Clinical Benefit is defined as the number of patients having a best overall tumour response of CR/PR or SD for ≥6 months.
  The Clinical Benefit rate is defined as the number of responders divided by the number in the Intention-to-treat (ITT) analysis set: responder=overall best response of complete response (CR)/partial response (PR) or stable disease (SD) for at least 6 months (calculated from the date of randomisation) as defined by RECIST criteria at any point prior to the data cut-off.
Time Frame: Every 8 weeks until progression or discontinuation
Measure: Number; unit: Ratio
Arm/Group | Cediranib 45 mg | Placebo
Number analyzed (Participants) | 31 | 31
Ratio | 0.419 | 0.419

5. Secondary Outcome: Duration of Clinical Benefit
Description: Number of days from date of clinical benefit to date of progression. Clinical benefit is defined as having a best overall tumour response of CR/PR or SD for ≥6 months.
Time Frame: Every 8 weeks until progression or discontinuation
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cediranib 45 mg | Placebo
Number analyzed (Participants) | 13 | 13
Days | 306.6 (104.2) | 343.8 (115.8)

ADVERSE EVENTS:
Arm/Group | Cediranib 45 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 15/31 | 4/31
Other Adverse Events (participants affected / at risk) | 29/31 | 30/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib 45 mg (N=31) | Placebo (N=31)
Intracardiac Thrombus (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Multi-Organ Failure (General disorders) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Weight Decreased (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Water Intoxication (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Convulsion (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 4 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib 45 mg (N=31) | Placebo (N=31)
Hypothyroidism (Endocrine disorders) | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 20 | 4
Constipation (Gastrointestinal disorders) | 11 | 4
Stomatitis (Gastrointestinal disorders) | 11 | 3
Vomiting (Gastrointestinal disorders) | 11 | 3
Nausea (Gastrointestinal disorders) | 10 | 8
Abdominal Pain (Gastrointestinal disorders) | 6 | 3
Dyspepsia (Gastrointestinal disorders) | 4 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 2
Dry Mouth (Gastrointestinal disorders) | 2 | 3
Oral Pain (Gastrointestinal disorders) | 3 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 2
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 1
Gingival Bleeding (Gastrointestinal disorders) | 2 | 1
Toothache (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 19 | 8
Asthenia (General disorders) | 6 | 0
Oedema Peripheral (General disorders) | 3 | 3
Pyrexia (General disorders) | 3 | 2
Chills (General disorders) | 2 | 1
Injection Site Pain (General disorders) | 1 | 2
Non-Cardiac Chest Pain (General disorders) | 2 | 0
Pain (General disorders) | 2 | 1
Urinary Tract Infection (Infections and infestations) | 4 | 2
Nasopharyngitis (Infections and infestations) | 1 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 2
Weight Decreased (Infections and infestations) | 6 | 0
Weight Increased (Infections and infestations) | 0 | 3
Anorexia (Metabolism and nutrition disorders) | 12 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 7
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 6 | 5
Bone Pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 3
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Headache (Nervous system disorders) | 11 | 7
Dizziness (Nervous system disorders) | 5 | 3
Dysgeusia (Nervous system disorders) | 5 | 0
Paraesthesia (Nervous system disorders) | 1 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 2
Somnolence (Nervous system disorders) | 2 | 2
Anxiety (Psychiatric disorders) | 1 | 3
Insomnia (Psychiatric disorders) | 1 | 2
Breast Pain (Reproductive system and breast disorders) | 1 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 11 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 4 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 | 0
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 16 | 6
Hot Flush (Vascular disorders) | 3 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a Study Site, or an investigator, requests permission to publish data from this study, any such publication (including oral presentations) is to be agreed with AstraZeneca prior to publication.